CLINICAL TRIAL: NCT03638830
Title: Randomized, Blind, Placebo-controlled Study to Evaluate Safety and Efficacy of Ftortiazinon in Combination With Maxipime®, in Comparison With Placebo in Combination With Maxipime®, in the Treatment of Patients With Complicated Urinary Tract Infections Caused by P. Aeruginosa
Brief Title: Safety and Efficacy Study of Ftortiazinon in the Treatment of Patients With Complicated Urinary Tract Infections Caused by P. Aeruginosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Acellena Contract Drug Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-FT-2018
Record Dates: First submitted 2018-08-07; First posted 2018-08-20 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Patients With Complicated Urinary Tract Infections Caused by P. Aeruginosa; Pseudomonas Aeruginosa; Pseudomonas Infections; Urinary Tract Infections
Keywords: Pseudomonas Aeruginosa; antibiotic resistance; factors of pathogenicity of bacteria; the system of secretion of type III pathogenic bacteria; Pseudomonas Infections; Urinary Tract Infections
MeSH Terms: conditions — Pseudomonas Infections; Urinary Tract Infections | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: randomized, blind, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: In order to minimize subjectivity, block randomization will be carried out in treatment groups without stratification in the center. Randomization will be carried out by the method of envelopes.
  To minimize the subjectivity of clinical study of the efficacy and safety of the drug "Ftortiazinon" will be conducted with the use of a placebo, which will not differ in appearance, shape, color, and will fully simulate the investigated product.
  To distribute the drug to patients, taking into account the need to observe the blinding, a special authorized person (an unblided research pharmacist) will be appointed in each medical organization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Ftortiazinon tablets 300 mg (FSBI "N.F. Gamaleya NRCEM" of the Ministry of Health of the Russian Federation)1/2 dose + placebo+ Maxipime®
  Interventions: Drug: Ftortiazinon (tablets 300 mg) 1/2 dose +placebo+ Maxipim
- Group 2 (Experimental): Ftortiazinon tablets 300 mg (FSBI "N.F. Gamaleya NRCEM" of the Ministry of Health of the Russian Federation) full dose + Maxipime®
  Interventions: Drug: Ftortiazinon (tablets 300 mg) full dose + Maxipim
- Group 3 (Placebo Comparator): placebo (like full dose) in combination with the drug Maxipime®
  Interventions: Other: placebo+Maxipim

INTERVENTIONS:
Drug: Ftortiazinon (tablets 300 mg) 1/2 dose +placebo+ Maxipim — Ftortiazinon tablets 300 mg (FSBI "N.F. Gamaleya NRCEM" of the Ministry of Health of the Russian Federation)+placebo
  Arms: Group 1
Drug: Ftortiazinon (tablets 300 mg) full dose + Maxipim — Ftortiazinon tablets 300 mg (FSBI "N.F. Gamaleya NRCEM" of the Ministry of Health of the Russian Federation)
  Arms: Group 2
Other: placebo+Maxipim — placebo
  Arms: Group 3

SUMMARY:
This study is planned to evaluate the safety and efficacy of the drug Ftortiazinon in combination with the drug Maxipime® in comparison with placebo in combination with the drug Maxipime® in the treatment of hospitalized adult patients with complicated urinary tract infections caused by P. aeruginosa.

DETAILED DESCRIPTION:
The study is divided into 2 phases.

The course of treatment will be single (course of therapy with the drug/placebo under study) for a group consisting of three cohorts, and also single for a group of phase 2 participants (770 patients in total) consisting of two cohorts groups. The recruitment of patients to the second phase will commence after the evaluation of the data on safety and efficiency by the expert commission within the framework of reviewing the amendment to the current Study Protocol. At the second phase, it is proposed to study the optimal dosage chosen based on the results of the first (search phase) study.

This study is aimed at evaluating the efficacy, safety and tolerability of the drug Ftortiazinon tablets 300 mg (FSBI "N.F. Gamaleya NRCEM" of the Ministry of Health of the Russian Federation) in combination with the drug Maxipime®, a powder for the preparation of a solution for intravenous and intramuscular administration of 1.0 g (Bristol-Myers Squibb, USA), in comparison with placebo in combination with the drug Maxipime®, a powder for the preparation of a solution for intravenous and intramuscular administration of 1.0 g (Bristol-Myers Squibb, USA), in the treatment of patients with complicated urinary tract infections (complicated UTIs) caused by P. aeruginosa.

FIRST PHASE (search phase) At this phase, the patients will take the drug Ftortiazinon tablets 300 mg (FSBI "N.F. Gamaleya NRCEM" of the Ministry of Health of the Russian Federation) in combination with the drug Maxipime®, a powder for the preparation of a solution for intravenous and intramuscular administration of 1.0 g (Bristol-Myers Squibb, USA).

According to the results of the screening of patients who have signed the Informed Consent Form, the patients are recruited in three groups with different doses of the drug. The total number of patients who received the drug or placebo will be at least 240 people according to the following scheme:

Group 1 (80 patients) - Ftortiazinon tablets 300 mg (FSBI "N.F. Gamaleya NRCEM" of the Ministry of Health of the Russian Federation) plus placebo. The drug is administered according to the following scheme on the first day: the first administration of Ftortiazinon 300 mg (1 tablet) plus placebo (1 tablet) 30 minutes after eating with lukewarm water, the second administration - 1 tablet (300 mg) after 12 hours, then within 6 days the drug is prescribed 1 tablet once a day plus 1 tablet of placebo (interval: 12 hours) 30 minutes after eating.

Group 2 (80 patients) - Ftortiazinon tablets 300 mg (FSBI "N.F. Gamaleya NRCEM" of the Ministry of Health of the Russian Federation). The drug is administered according to the following scheme on the first day: the first administration of 600 mg (2 tablets) 30 minutes after eating with lukewarm water, the second administration - 1 tablet (300 mg) after 12 hours, then within 6 days the drug is prescribed 1 tablet twice a day at intervals of 12 hours.

Group 3 (80 patients) - placebo in combination with the drug Maxipime®, a powder for the preparation of a solution for intravenous and intramuscular administration of 1.0 g (Bristol-Myers Squibb, USA). The drug is administered according to the following scheme on the first day: the first administration of 2 tablets 30 minutes after eating with lukewarm water, the second administration - 1 tablet after 12 hours, then within 6 days the drug is prescribed 1 tablet twice a day at intervals of 12 hours 30 minutes after eating.

For all groups: Maxipime®, a powder for the preparation of a solution for intravenous and intramuscular administration of 1.0 g (Bristol-Myers Squibb, USA). The drug is administered according to the following scheme: the drug with a dosage of 1.0 g is dissolved in 2.4 ml of sterile water for injection or 0.9% sodium chloride solution, or 0.5-1% lidocaine hydrochloride solution; then injected deep into the muscle, into the upper outer quadrant of the buttocks after pre-aspiration every 12 hours for 7 days*.

SECOND PHASE (confirmation phase) The transition to this phase of the study to assess efficacy and safety of the drug Ftortiazinon will be carried out after selecting the optimal dosage according to the results of the first (confirmation phase) study.

This transition will be carried out by making a corresponding amendment to the Study Protocol with the provision of data confirming the efficacy and safety of the selected therapeutic scheme.

The assessment will be conducted according to the results of the 21-day surveillance for patients after completion of therapy with a drug/placebo.

Group 1 patients will take the drug Ftortiazinon tablets 300 mg (FSBI "N.F. Gamaleya NRCEM" of the Ministry of Health of the Russian Federation) in combination with the drug Maxipime®, a powder for the preparation of a solution for intravenous and intramuscular administration of 1.0 g (Bristol-Myers Squibb, USA) in accordance with the dosage regimen selected at the first phase.

Maxipime® is a powder for the preparation of a solution for intravenous and intramuscular administration of 1.0 g (Bristol-Myers Squibb, USA). It is administered according to the following scheme: the drug with a dosage of 1.0 g is dissolved in 2.4 ml of sterile water for injection or 0.9% sodium chloride solution, or 0.5-1% lidocaine hydrochloride solution; then injected deep into the muscle, into the upper outer quadrant of the buttocks after pre-aspiration every 12 hours for 7 days.

Group 2 patients will take placebo in combination with the drug Maxipime®, a powder for the preparation of a solution for intravenous and intramuscular administration of 1.0 g (Bristol-Myers Squibb, USA). Placebo is taken according to the scheme corresponding to those chosen at the first phase.

Maxipime® is a powder for the preparation of a solution for intravenous and intramuscular administration of 1.0 g (Bristol-Myers Squibb, USA). It is administered according to the following scheme: the drug with a dosage of 1.0 g is dissolved in 2.4 ml of sterile water for injection or 0.9% sodium chloride solution, or 0.5-1% lidocaine hydrochloride solution; then injected deep into the muscle, into the upper outer quadrant of the buttocks after pre-aspiration every 12 hours for 7 days.

Administration/injection of drugs Ftortiazinon/placebo and Maxipime® should be carried out simultaneously, preferably in one and the same time every day. Let the administration of Ftortiazinon/placebo will be for 30 min after administration of the drug Maxipime®.

The duration of therapy with Maxipime® will be 7 calendar days; however, if the patient has no positive dynamics in the evaluation of clinical symptoms of complicated UTIs, there is an increase in uropathogen in the urine culture obtained on Visit 2, and the duration of therapy can be increased to a total of 14 calendar days.

ELIGIBILITY:
Inclusion Criteria:

* 1. The ability to understand the requirements of the study participants, to give written consent to participate in the study (including the use and transfer of information about the patient's health related to the study) and the implementation of the procedures provided by the Study Protocol.

  2. Availability of the patient's written consent to participate in the study according to the current legislation.

  3. Male or female participants must be ≥18 and ≤80 years of age. 4. It is expected that patient's treatment of complicated UTI will require hospitalization and the use of antibiotic therapy.

  5. Suspected or documented complicated UTI as defined below and subject to the mandatory presence of one or more of the risks associated with the complicated UTI listed below:

Complicated urinary tract infection (complicated UTI):

• presence of at least 2 of the following signs or symptoms:

* chills, tremors, or body temperature increases associated with fever (body temperature of 38ºC) (fever documented by a medical professional within 24 hours prior to screening);
* nausea or vomiting within 24 hours prior to screening;
* dysuria, frequent urination or urgent need to urinate;
* pain in the lower abdomen;
* acute pain in the side (occurred within 7 days prior to randomization) or pain in the region of the rib-vertebral angle during physical examination.

  • leukocyturia in a urine sample (presence of at least one of the following signs):
* positive reaction to leukocyte esterase based on the results of the common urine examination;
* number of leukocytes ≥ 10 cells/mm3 in non-centrifuged urine sample;
* number of leukocytes ≥ 10 cells / per HPF in the urine sediment. 6. At least one of the following associated risks: • periodic bladder catheterization or the presence of a permanent bladder catheter, ureters (ureter stent), kidneys (nephrostoma) (catheters installed more than 24 hours prior to screening should be removed or replaced prior to collection of an urine sample for analysis and sowing, unless removal or replacement is considered unsafe or contraindicated);

  * presence of known functional or anatomical abnormalities in the urinary system, including malformations, neurogenic bladder, presence of residual urine volume ≥ 100 ml, stricture after surgery and/or malformations of the urinary tract, separate drainage of the kidney and/or bilateral nephrostomy tubes;
  * complete or partial obstructive uropathy (e.g. nephrolithiasis, tumor, fibrosis, urethral stricture, cystolithiasis) that is expected to be subjected to therapeutic or surgical treatment during treatment with the drug under study (until the end of therapy);
  * azotemia defined as blood urea nitrogen level (BUN) > 20 mg/dl, blood urea level > 42.8 mg/dl, or serum creatinine > 1.4 mg/dl due to known kidney disease in anamnesis;
  * chronic urinary retention in men, e.g. due to the previously diagnosed benign prostatic hypertrophy.

    7. Obtaining the patient's initial urine sample for sowing within 24 hours before randomization (patients can be randomized in this study and start therapy with the drug under study before the results of the initial urine culture become known to the researcher).

    8. A reasonable assumption that any installed urinary device (e.g., nephrostomy catheter, permanent stents) will be surgically removed or replaced before or within 24 hours of randomization (temporary catheters that were installed more than 24 hours before screening should be removed or replaced before urine sample collection for analysis and sowing).

    9. Recurrent complicated urinary tract infection within 12 months before the study (presence of complicated urinary tract infection in anamnesis with a frequency of more than twice per year).

    10. Suspected infection caused by multiresistant strains of P. aeruginosa, inefficiency of previous treatment.

    11. High risk of complicated UTI caused by P. aeruginosa (e.g. pseudomonal complicated UTI in anamnesis, therapy of 20 mg or more with prednisone or equivalent steroid and other risk factors that are taken into account by the researcher.

    12. Prognostic life expectancy of the patient with effective antibiotic therapy and proper maintenance treatment is estimated by the researcher to be at least 6 months.

    13. Women who capable of childbirth (i.e. not in menopause and not surgically sterilized) should have a negative pregnancy test result before randomization. Participants in the study who are capable of procreation, or sexual partners of participants who are capable of childbirth, should agree to the continued use of a highly effective method of contraception from the beginning of screening to the end of the study (medical and pedagogical observations) (highly effective methods of contraception include hormonal implants, plasters, injectable hormones, oral hormonal contraceptives, intrauterine systems, approved cervical ring, prior bilateral ovariectomy, prior hysterectomy, previous bilateral tubal ligation, true abstinence from sexual activity (if confirmed by the researcher), or vasectomy with a partner.

    14. Male participants of the study will need to use condoms with spermicide during sexual intercourse during screening up to the end of the study in case of possible and even existing pregnancy of the sexual partner.

Exclusion Criteria:

* 1. Presence of any known or suspected disease, or condition that may distort the assessment effectiveness, including, but not limited to, the following:

  * perinephral abscess;
  * corticomedullary kidney abscess;
  * any history of pelvic or urinary tract injury within 30 days prior to the study;
  * polycystic kidney disease;
  * chronic vesicoureteral reflux;
  * prior or planned kidney transplantation;
  * dialysis patients, including those under hemodialysis, peritoneal dialysis or continuous venovenous hemofiltration (CVVH);
  * previous or planned cystectomy or surgery on the loop of ileum;
  * presence of a known or suspected infection that is caused by fungi (e.g. candiduria) or mycobacteria (e.g. urogenital tuberculosis).

    2. Presence of suspected or confirmed acute bacterial prostatitis, orchitis, epididymitis or chronic bacterial prostatitis determined by anamnesis and/or general medical examination.

    3. Macrogematuria requiring treatment other than administration of the drug under study or removal, or replacement of the urinary catheter.

    4. Surgery on the urinary tract within 7 days before randomization, or surgery on the urinary tract planned during the period of study (except surgical intervention necessary to remove the obstruction or placement of the stent or holding of a nephrostomy until the end of treatment (medical and pedagogical observations).

    5. Renal function in screening evaluated by creatinine clearance as < 50 ml / min using the Cocroft-Gault formula and serum creatinine values obtained in a local laboratory.

    6. Source of infection diagnosed within 7 days prior to randomization with known extra-renal origin, such as endocarditis, osteomyelitis, abscess, burn urinary tract infection; meningitis or pneumonia.

    7. Any signs of sepsis, including shock or deep arterial hypotension, which is defined as SBP < 90 mm Hg or a pressure reduction of > 40 mm Hg from the initial level (if known) not reacting to the load with a liquid.

    8. Pregnant or breastfeeding women. 9. Established epileptic syndrome requiring ongoing treatment with an anticonvulsant drug, which will not allow the patient to comply with the treatment regimen according to the Study Protocol. Patients with a history of epilepsy or those receiving stable therapy (i.e. unchanged therapy for 30 days) with a well-controlled epileptic syndrome (i.e. with no recurrence within the last 30 days) may be considered for admission to the study.

    10. Treatment with antitumor chemotherapeutic drugs, treatment with immunosuppressive therapy for transplantation, or drugs preventing rejection of the transplant within 30 days prior to randomization.

    11. Signs of severe disease or liver dysfunction, including confirmed viral hepatitis or hepatic encephalopathy.

    12. AST or ALT > 3 x ULN (upper limit of normal) or total bilirubin > 1.5 x ULN at screening.

    13. Administration of any long-acting systemic antibiotic (i.e. with a frequency of less than once per day) for less than 12 hours prior to randomization.

However, the following patients may be included:

• who have received antimicrobial therapy for > 24 hours and have not responded to treatment (i.e. signs and symptoms have worsened) and have documented complicated UTIs caused by pathogen microorganisms resistant to previous therapy;

* who developed signs and symptoms of complicated UTI in the administration of systemic antibiotics for other indications, including antimicrobial prophylaxis against recurrent UTI;
* who received short-acting systemic antibiotic therapy (i.e. with frequency of administration more than once per day) for 24 hours before randomization, but not less than 12 hours prior to randomization.

  14. Need for additional systemic antimicrobial therapy at the time of randomization (including antibiotic, antifungal therapy), other than treatment with the drug under study, except for a single oral administration of any antifungal drug for the treatment of vaginal candidiasis.

  15. Likelihood of the need for an antibiotic to prevent complicated UTI during patient participation in the study (from randomization to medical and pedagogical observations).

  16. Impossibility of removal or replacement of temporary catheters installed in more than 24 hours prior to the screening from the perspective of evaluating the safety of the patient or presence of contraindications to manipulation (temporary catheters installed more than 24 hours prior to the screening should be removed or replaced prior to collecting the urine sample for analysis and sowing).

  17. History of HIV infection. 18. Presence of significant immunodeficiency or immune deficiency, including hematologic malignant disease, bone marrow transplantation or receiving immunosuppressive therapy, such as chemotherapy for cancer, administration of drugs to prevent graft rejection and long-term use of systemic corticosteroids (equivalent to the use of prednisone or equivalent systemic drug at a dose ≥ 20 mg/day for ≥ 2 weeks).

  19. Presence of neutropenia (absolute number of neutrophils < 1000/mm3) based on the results of the screening analysis in the central laboratory.

  20. Presence of thrombocytopenia (especially in patients diagnosed with disseminated intravascular coagulation or risk of serious bleeding) 50,000 platelets/mm3 confirmed on the basis of indicators obtained in the central laboratory during screening.

  21. Lactose intolerance, lactose deficiency or glucose-galactose absorption, severe hypersensitivity or allergic reaction to β-lactam antibiotics, L-arginine, local anesthetics, antiarrhythmics or to the components of the drug in anamnesis.

  22. Presence of any contraindications to the use of β-lactam antibiotics (cephalosporins, penicillins, carbapenems or monobactams), to administration of auxiliary substances that are part of the relevant dosage forms.

  23. Participation in another clinical trial using the drug or device under study for the last 90 days prior to randomization.

  24. Inability or unwillingness to comply with the requirements of the Study Protocol.

  25. Any patients previously randomized into this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 777 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
clinical cure and microbiological eradication | through the whole study, an average of 90 days
  proportion of patients with overall positive effect

SECONDARY OUTCOMES:
proportion of patients with clinical cure response | through the whole study, an average of 90 days
  proportion of patients with clinical cure response in the patient population treated with the drugs specified in the Study Protocol, i.e. corresponding to the MITT criterion, in the group of patients with the isolated pathogen P. aeruginosa in urine at baseline, i.e. corresponding to the m-MITT criterion, patient population suitable for clinical evaluation (CE), and patient population suitable for microbiological evaluation (ME)
proportion of patients with response in the form of microbiological eradication | through the whole study, an average of 90 days
  proportion of patients with response in the form of microbiological eradication in the m-MITT and ME populations during medical and pedagogical observations;
microbiological eradication | day 7
  microbiological eradication for each selected pathogen in the m-MITT and ME populations during medical observations
number of patients with treatment response as clinical cure | day 7
  relative number of patients with treatment response as clinical cure in the MITT and m-MITT populations
Number of Participants With Adverse Events | through the whole study, an average of 90 days
  Determination of Number of Participants With Adverse Events
Number of Participants With Serious Adverse Events | through the whole study, an average of 90 days
  Determination of Number of Participants With Serious Adverse Events
Number of Participants with Solicited Local and Systemic Adverse Events | through the whole study, an average of 90 days
  Determination of Number of Participants with Solicited Local and Systemic Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Victor Shunkov, MD, PhD, Principal Investigator — Road Clinical Hospital of Open Joint Stock Company "Russian Railways; Alexander Shvets, MD, Principal Investigator — Saint-Petersburg Clinical Hospital of the Russian Academy of Sciences; Dmitry Gorelov, MD, Principal Investigator — Scientific and Research Center "Eco-Safety"; Lyudmila Kulagina, MD, Principal Investigator — Republican Clinical Hospital of the Ministry of Health of the Republic of Tatarstan; Elena Matevosyan, MD, Principal Investigator — Vsevolozhsk Clinical Interdistrict Hospital; Maria Mozheyko, MD, Principal Investigator — Yaroslavl Regional Clinical Hospital for Military Veterans; Lev Sinelnikov, MD, Principal Investigator — S.M. Kirov Military Medical Academy; Maksim Bushara, MD, Principal Investigator — Baltic Medicine; Ashot Yesayan, MD, Principal Investigator — Saint-Petersburg State Budgetary Healthcare Institution "City Clinical Hospital No. 31"; Alexander Mangushlo, MD, Principal Investigator — St. Petersburg state budgetary institution of health care " City hospital № 26"; Andrey Gorelov, MD, Principal Investigator — St. Petersburg state budgetary institution of health care " city Pokrovskaya hospital"; Grigory Arutunov, MD, Principal Investigator — Pirogov Russian National Research Medical University; Ivan Palagin, MD, Principal Investigator — Smolensk regional clinical hospital; Igor Shormanov, MD, Principal Investigator — State Autonomous healthcare institution of Yaroslavl region Clinical hospital № 9
Locations (5):
- Russia (5):
  - Road Clinical Hospital of Open Joint Stock Company "Russian Railways, Saint Petersburg, Sankt-Peterburg
  - St. Petersburg state budgetary institution of health care " City hospital № 26", Saint Petersburg, Sankt-Peterburg
  - Baltic Medicine, Saint Petersburg
  - Scientific and Research Center "Eco-Safety", Saint Petersburg
  - Vsevolozhsk Clinical Interdistrict Hospital, Vsevolozhsk

IPD SHARING:
Plan to Share IPD: No